CLINICAL TRIAL: NCT02141906
Title: A Pilot Study of "OncozeneTM" Microspheres for Intra-arterial Delivery of Doxorubicin for the Treatment of Patients With Unresectable Hepatocellular Cancer
Brief Title: A Pilot Study of "OncozeneTM" Microspheres for Intra-arterial Delivery of Doxorubicin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Muhammad Beg, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 012014-079
Record Dates: First submitted 2014-04-30; First posted 2014-05-20 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncozene-DEB-TACE (Experimental): Screening Visit (procedures should be done within 28 days of treatment day):
  Study visit assessments will be performed prior to Oncozene-DEB-TACE delivery (except pharmacokinetic blood draw).
  Labs may be done within 3 days of the procedure. All visits can be completed +/- 10 days of planned visit day
  Follow up after completion of treatment every 4-6 weeks:
  Interventions: Other: Oncozene-DEB-TACE

INTERVENTIONS:
Other: Oncozene-DEB-TACE — ONCOZENE microspheres are the newly available microspheres for DEB-TACE. It appears (based on the preliminary bench tests) that these microspheres may allow more efficient drug loading, and slow elution and equivalent vascular occlusion(12). In this pilot study, we aim to assess the safety of these microspheres when used for chemoembolization of unresectable hepatocellular carcinoma.
  Other Names: Oncozene microspheres for Doxurubicin delivery

SUMMARY:
This is a pilot study of Onconzene Microspheres for intra-arterial delivery of doxorubicin for the treatement of patients with unresectable hepatocellular cancer.

DETAILED DESCRIPTION:
The study will evaluate the safety and tolerability of doxorubicin loaded ONCOZENE microspheres chemoemobilization for the treatment of unresectable hepatocellular carcinoma.

The study will also describe the overall response rates of lesions with Oncozene-DEB-TACE(Trans-arterial chemoemobilization) per modified RECIST criteria (Response Evaluation Criteria in Solid Tumors).

Determine progression free survival (PFS) and overall survival (OS) following Oncozene-DEB-TACE (Trans-arterial chemoemobilization)

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Hepatocellular carcinoma confirmed by at least one of the following: a) histological confirmation; b) imaging results consistent with cirrhosis and at least one solid liver lesion of >2cm with early enhancement and delayed washout (AASLD criteria for diagnosis of HCC); c) Alpha fetoprotein level >400ng/mL and evidence of at least one solid liver lesion >2cm, regardless of specific imaging characteristics on MRI.
* Tumor not suitable for resection at the time of study entry. (Transplant eligible patients are allowed)
* Age ≥ 18 years.
* Performance status ECOG PS 0-1 (Eastern Cooperative Oncology Group Performance Status).
* Child Pugh Score A only
* Adequate organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mcL (Measurement and Calibration Lab)
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 75,000/mcl
  * total bilirubin ≤ 3.0
  * AST (Aspartate Aminotransferase)(SGOT)/ALT (Alanine Aminotransferase)(SPGT) ≤ 5 X institutional upper limit of normal
  * creatinine ≤ 2.0
  * INR (International Normalized Ratio) ≤ 1.8
  * Albumin ≥ 2.8
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* Has not undergone a hysterectomy or bilateral oophorectomy
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Absence of occlusive thrombus in the main portal vein
* Life expectancy of at least 6 months
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks prior to entering the study or those with residual treatment related toxicity of greater than grade 1 not addressed in inclusion criteria.
* Any concurrent therapy for HCC including concurrent investigational agents.
* Subjects with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to doxorubicin or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Child-Pugh status B or C
* Encephalopathy no adequately controlled medically
* Known cardiac ejection fraction <50%
* Tumor involving >50% of the liver
* Infiltrative form of HCC on imaging; If there is at least one measurable lesion per mRECIST criteria and otherwise patient is eligible for the study, the patient can be enrolled.
* Extensive extrahepatic spread of hepatocellular carcinoma. Patients with limited metastatic disease may be enrolled as defined as

  * lymph node disease
  * pulmonary nodules <5 mm in size
  * 1-3 bone metastases
* Active gastrointestinal bleeding
* Evidence of uncontrollable bleeding diathesis
* Any contra-indication to angiography
* Any known contra-indication to chemoembolization according to the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Response | (Oncozene-DEB-TACE): TACE 1 Day 22-28, TACE 2-6 Day 22-28, Follow up after completion of treatemtent every 4-6 weeks up to 36 weeks.
  Treatement response will be measured using modified RECIST assessment for hepatocellular cancer. Patients will undergo a maximum of 3 treatments each, at least 4 weeks apart unless there is a complete response as per mRECIST criteria (no enhancing tumor on subsequent CT or MRI scan)

SECONDARY OUTCOMES:
Progression | (Oncozene-DEB-TACE): TACE 1 Day 22-28, TACE 2-6 Day 22-28, Follow up after completion of treatemtent every 4-6 weeks up to 36 weeks.
  Treated lesion will be evaluated for progression. Progression will be defined according to the mRECIST criteria (Response Evaluation Criteria in Solid Tumors).Patients will undergo a maximum of 3 treatments each, at least 4 weeks apart unless there is a complete response as per mRECIST criteria (no enhancing tumor on subsequent CT or MRI scan)
  .

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Beg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No